

VSTAT COVID: Vadadustat Study Targeting ARDS Therapy in COVID and VSTAT-LoTuS: A Long- Term Follow Up Study of COVID-19 Patients treated with either vadadustat or placebo.

NCT04478071

Version Date: 01/20/2022

# CONSENT TO TAKE PART IN RESEARCH

HSC-MS-20-0395

# **Simple Study Title:**

VSTAT-LoTuS

# **Full Study Title:**

VSTAT COVID: Vadadustat Study Targeting ARDS Therapy in COVID and VSTAT-LoTuS: A Long-Term Follow Up Study of COVID-19 Patients treated with either vadadustat or placebo.

# **Study Sponsor:**

McGovern Medical School at UTHealth

# **Principal Investigator:**

Bentley J. Bobrow MD

# **Study Contact:**

# **Purpose:**

The purpose of this study is to assess how well an oral drug called vadadustat given once a day for 14 days works for the prevention and treatment of acute respiratory distress syndrome (ARDS) in patients hospitalized with COVID-19 infection. **This is a voluntary study** and if you choose to participate, you will be asked to sign this consent form that you agree to be part of the study. If you have any questions at any time or need clarification on anything, or would like a language translator, please ask

The goal of this study is to see how well vadadustat the drug to be tested, works at preventing and treating people with COVID-19 infection, your current condition. This drug is not yet approved by the Food and Drug Administration (FDA); therefore, it is called an investigational drug. The study is funded through Akebia Therapeutics Inc. located in Cambridge, MA. Akebia is paying UTHealth for their work on this study. The Department of Defense (DoD) is also supporting this study.

A description of this clinical trial is available on <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>, as required by law. Your name or any personal information will not be publicly available. After the study has ended, the website will include a summary of the results. You can search this website at any time.

In this study, a drug called vadadustat or placebo will be given to you by mouth each day with the goal of decreasing inflammation in your lungs and to reduce the chance you may need a ventilator due to the COVID-19 infection. The total amount of time you will be in this study is 28 days. This will include the time you are in the hospital and then after you go home. On day 28 you will be contacted by the research team for follow up. If you agree and are able to take part in this study you will undergo the following procedures:

Contact Name: Revised 12/23/2021

IRB NUMBER: HSC-MS-20-0395

- As part of the study procedure, a small sample of blood (10 ml) will be drawn prior to starting the drug, then again on day 7 and on day 14.
- The study drug, vadadustat or a placebo, will be administered every day for 14 days by mouth or if you are placed on a ventilator through a nasogastric tube that your doctor will position. You will be given six small tablets (each about the size of a baby aspirin), a total of 900 mg once a day.
- You will be followed carefully and assessed to see whether your COVID-19 infection worsens or improves and how quickly that happens.

#### Risks:

There are potential risks involved with this study that are described in this document. There are both risks and benefits to taking part in this study. It is important for you to think carefully about these as you make your decision.

Some known risks include:

- If you choose to take part in this study, there is a risk that the vadadustat may not be helpful in treating your condition.
- There is a small risk of having a bruise, bleeding or discomfort at the site of the needle stick for drawing blood, although we will be taking this blood at the same time as your other blood tests are performed, so this will be unlikely.
- The most commonly known side effect of vadadustat is gastrointestinal upset such as nausea and vomiting which is usually mild.
- Patients who have COVID-19 are at increased risk for abnormal blood clotting. While this has not been detected in clinical studies, there is a theoretical risk that taking vadadustat may increase the risk of abnormal blood clotting. If your physician deems appropriate, you may receive a blood thinner.
- As we will need to collect some information about your healthcare and blood test results, there are possible risks from loss of confidentiality that may arise from taking part in the study. Please be assured that we will take every precaution to protect your health information in compliance with all hospital, state, and federal regulations and we are committed to preventing this from happening.

You will also be monitored for any serious adverse effects (SAEs) by your physician and the UTHealth Research Team.

#### **Benefits:**

We are doing this study because UTHealth physician-scientists believe that there is a strong chance that the drug vadadustat given to patients with COVID-19 could help prevent and/or treat acute respiratory distress syndrome (ARDS) which occurs when the lungs become inflamed and cannot function properly. We also are doing this study because we believe that some very important information will be discovered which may help the medical team treating you. However, even if this drug does not ultimately help patients with COVID-19, the information from this study may show us how to better help future patients who are receiving treatment for ARDS.

Alternatives: You may choose not to take part in this study. Participation in this research study is completely voluntary. You may also choose to stop the research study at any time. Your decision will not in any way affect the clinical care you receive. If you are interested in participating, please continue to read below.

Who is being asked to take part in this study?

Contact Name: Revised 12/23/2021



You are being asked to take part in this research study because you have COVID-19 and are at risk for developing worsening acute respiratory distress syndrome (ARDS). This study is being conducted by physician scientists at UTHealth for patients in the Memorial Hermann Health and Harris Health System. Up to 650 adults will take part in the study.

# What will happen if I take part in this study?

You agree to be part of the study to treat ARDS due to the COVID-19. As part of the study procedure, small samples of blood (10 ml) will be drawn prior to the drug delivery and urine will be collected at time of enrollment, day 7 and at day 14. Blood and urine are being collected for analysis of organ and cell function. The study drug, vadadustat or placebo, will be administered every day for 14 days by mouth or if needed, through a nasogastric tube.

# If randomized to a treatment:

If you agree to take part in this study you will be randomized (similar to flipping a coin) to receive either the study drug vadadustat or the placebo (a tablet that contains no active ingredient). It is not known whether vadadustat will be of benefit. For this reason, some study participants must receive a placebo. This will allow a careful comparison to study the benefits and side effects of the investigational drug. There is a 50% chance you will receive vadadustat and a 50% chance that you will receive placebo. Neither you nor your doctor will know if you are receiving vadadustat or placebo, as both will look the same.

Exams, tests, and procedures, including but not limited to blood tests, need to be done as part of this study to monitor your safety and health, but may not be included in the usual care. We will use them to carefully follow the effects of the study treatment, including preventing and managing side effects.

# How long will you be in the study?

If you agree to take part, your participation will last for 14 days (hospitalization) and 14 days follow-up. You will receive a phone follow-up call after you go home on day 28 from when you first came to the hospital.

Additionally there is an opportunity to participate in an extended follow up period to determine the impact of COVID-19 and the trial on your health. If you choose to participate in this portion of the study you will be asked to:

- return to the clinic at 6, 12 and 24 months and during each visit:
- complete a quality of life questionnaire
- complete a cognitive questionnaire
- provide a blood sample (10 ml)
- provide a urine sample (10 ml)
- a nurse will perform a pulmonary function test and a doctor will perform a lung ultrasound to see how well your lungs are working, in addition to an ultrasound to see how your heart is working

If you would like to participate in the extended follow up, please check the box and initial below under the signature line.



# What choices do you have other than this study?

Your options are to participate in the study or not to participate in this study either way you will still be treated. You may decide to stop taking part in the study at any time. To withdraw from the study, please contact

Your doctor or the UTHealth Research Team can stop the study at any time. Your doctor or the UTHealth Research Team may stop your participation in the study if:

- your condition worsens
- the study is stopped
- the study drug is no longer available
- you do not meet all the requirements of the study,
- or the study is not in your best interest.

If your participation in the study is stopped, your doctor will discuss other options for your treatment. If you stop participating in this study, the information already collected about you will still be used in the data analysis. However, no further information will be collected without your permission.

While taking part in this study, the study team will notify you of new information that may become available and could affect your willingness to stay in the study.

Research participation is voluntary. Vaccines do exist but are not a cure and many people have not been able to receive vaccinations. COVID-19 ARDS has significant morbidity and mortality for high risk patient populations.

# What happens if you are injured during the study?

In the event of injury resulting from this research, UTHealth, Memorial Hermann System and/or the Harris Health system (Lyndon B. Johnson Hospital) are not able to offer financial compensation nor to absorb the costs of medical treatment. However, necessary facilities, emergency treatment and professional services will be available to you, just as they are to the general community. If you are injured or have any harmful effects during the course of the research study, treatment will be available to you. You or your insurance company will be billed for any treatment. You should report any such injury to You will not give up any of your legal rights by signing this consent form.

DoD will not provide compensation for any injury occurring during the study. DoD does not have a mechanism to provide compensation for study-related injury.

If you are inured, please report to the PI (Bentley Bobrow, MD at ) and to the Committee for the Protection of Human Subjects at Su signing this consent form.

# What are the costs of taking part in this study?

If you decide to take part in this research study, you will not incur any additional costs.

Upon completion of the D28 follow up call, a \$50 gift card will be mailed to you as a small token of appreciation.

If you choose to participate in the extended follow up, you will receive a \$100 gift card for each completed follow up visit. Parking and travel expenses will also be covered.

Contact Name: Revised 12/23/2021



The UTHealth will pay for the special tests and examinations that are required by this study and not otherwise part of your standard medical care.

However, many of the tests, procedures, and exams you will receive are believed to be part of standard medical care, and may or may not be covered by your medical insurance. If your medical insurance does not pay for your care you will be responsible for the cost of the medical care related to your condition including laboratory tests, deductibles, co-payments, physician and clinic fees, hospitalization and procedures.

| If you receive a bill that you believe is related to your taking part in this research study, please |
|---|
| contact: |

# How will privacy and confidentiality be protected?

Your privacy is important and your participation in this study will be kept confidential. However, absolute confidentiality cannot be guaranteed.

If you sign this document, you give permission to UTHealth, Memorial Hermann Healthcare System and/or Harris Health system to use and disclose (release) your health information. The health information that we may use or disclose for this research includes all information in a medical record, results of physical examinations, medical history, lab tests, or certain health information indicating or relating to a particular condition. Please understand that health information used and disclosed may include information relating to HIV infection, drug abuse, alcohol abuse, behavioral health, and psychiatric care.

If you sign this document, you give permission to UTHealth and/or Memorial Hermann Health System, and/or Harris Health System to use and disclose (release) your health information. Representatives of the organizations listed below will see your name and other personal identifiers when they review your research records and medical records for the purposes of verifying study data:

- Representatives of UTHealth and/or Memorial Hermann Health System and/or Harris Health System
- Representatives from the U.S.Food and Drug Administration (FDA)
- IQVIA
- AKEBIA
- The Department of Defense (DoD)
- Representatives of the sponsor for this research including contract research organizations
- Members of the Data and Safety Monitoring Boards (an independent group of experts that reviews this study's data to make sure participants are safe and re research data is reliable)
- Companies engaged with the UTHealth for the commercialization of the results of the research study

| Name of Provider | Address of Provider | Fax Number | of Provider |
|---|---|---|---|
| whom can you contact if you f you have questions at any times study team to discuss problem uestions about the research. | name and medical record number will ady. After we remove all identifiers, to with other researchers without you have questions about the study? me about this research study, please as he will be glad to arms, report injuries, voice concerns, of the of Human Subjects at the University | he information or<br>r additional info<br>e feel free to conswer your quest<br>otain information | or samples may be rmed consent. Intact the Dr. Bent ions. You can contain addition to ask |
| eviewed this research study. Yubject, and to discuss any conce | You may contact them for any questerns, comments, or complaints about | • | r rights as a res <u>ea</u> |
| sign below only if you understal art in this research study. You | You may contact them for any ques | taking part in a r<br>at the research ar<br>en answered. If y | r rights as a research study at |
| sign below only if you understal art in this research study. You | You may contact them for any questerns, comments, or complaints about and the information given to you about a sure that all your questions have be | taking part in a r<br>at the research ar<br>en answered. If y | r rights as a research study at |
| art in this research study. You understa art in this research study, a cop | You may contact them for any questerns, comments, or complaints about and the information given to you about a sure that all your questions have been of this signed consent form will be | taking part in a r<br>t the research ar<br>en answered. If y<br>given to you. | r rights as a research study at an at a research study at a resear |

Please check this box and initial if you would like to participate in the extended follow up.

